CLINICAL TRIAL: NCT03679338
Title: Prospective Evaluation of the Ablation Therapy With Bipolar Radio Frequency for Nonresectable Bile Duct Cancer
Acronym: RFA-BILIAIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFA-BILIAIRE-IPC 2016-003
Record Dates: First submitted 2017-11-14; First posted 2018-09-20 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Nonresectable Bile Duct Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation Therapy With Bipolar Radio Frequency (Other)
  Interventions: Device: Ablation Therapy

INTERVENTIONS:
Device: Ablation Therapy — Ablation Therapy With Bipolar Radio frequency

SUMMARY:
90 % of the patients with bile duct cancer are not justifiable of a surgical resection with curative aim for oncologic reasons ( metastatic extensions), for reasons of resectability (canalar extension, vascular) or still for surgically reasons (age, comorbidity).

The palliative care of these patients consists at first in assuring an effective biliary drainage, infectious complications being one of the main causes of death. The biliary drainage allows to improve the survival of these patients. It bases by the implementation, by the endoscopic or percutaneous way of biliary, generally metallic prosthesis the duration of average permeability of which is of approximately 6 months.

The standard oncologic treatment is the administration of a chemotherapy exclusive or associated with a radiotherapy. The radiotherapy and the radio chemotherapy did not show efficiency on the survival superior to the exclusive biliary drainage. The first-line exclusive chemotherapy bases on the gemcitabine-cisplatin association with a median survival of 11,6 months. No study allows to justify the administration of a chemotherapy of the second line.

Thus the preservation of the permeability of the biliary ways is today, the most important factor to improve the survival of these patients. Therefore, the addition of a treatment allowing to obtain a local tumoral response to the insertion of biliary prosthesis would allow to increase the duration of permeability of the biliary prosthesis and would limit the local evolution.

Endoductal destruction tumoral technics were thus developed in this indication:

1. Dynamic phototherapy which demonstrated, during preliminary studies, a certain efficiency both on the tumoral response estimated on the improvement of the tumoral stenosis as on the survival in case of cholangiocarcinoma bile ducts not resectables. However, the improvement of the survival was not confirmed by wider randomized studies. A study randomized of phase III was interrupted prematurely because of a survival decreased in the experimental arm.
2. The radium therapy and the brachytherapy were estimated in this indication with results interesting on series limited in size, but is not used in routine because of its cost and of technics difficulties.

Ablation therapy technics (radio frequency, microwaves, radium therapy) percutaneous by radiological or surgical way proved their efficiency for the treatment of hepatocarcinoma and liver metastasis.

The hepatic radio frequency was estimated, during trials of phases II, for peripheral cholangiocarcinoma intra hepatic (developed at a distance main bile ducts) with interesting tumoral rates of necrosis.

However, the direct percutaneous access of the cholangiocarcinoma of the biliary ways is not practicable because of the risk of iatrogenic biliary fistula.

Therefore, systems allowing to realize ablation therapy by endoductal radio frequency are from now on available. It is miniaturized bipolar probes which are inserted into bile ducts by reactionary way (retrograde cholangiography), or anterograde percutaneous.

Two systems (Habib ®, ELLRA ®) are at present available and were estimated during in vitro and in vivo studies, to the animal and in man.

The purposes of this study are to estimate the feasibility, the efficiency and the morbidity of the biliary radio frequency for the treatment of the extra hepatic cholangiocarcinoma non resectable (resection or transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Bile duct cancer nonresectable
* Type I, II ou III of Bismuth classification with cholangio-MRI and/or endoscopic cholangiography
* Laboratory values : prothrombin time ≥ 50%, platelets ≥ 50 000, aPTT < 3 (Authorized transfusions)
* Written informed consent,
* Affiliation to Social Security System.

Exclusion Criteria:

* Intra-pancreatic mass and/or Wirsung dilation,
* Bile duct cancer,
* Visceral metastasis (extrahepatic),
* Initial metallic prosthesis,
* Woman pregnant or susceptible to the being,
* Patients deprived of liberty or placed Under the authority of a tutor,
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Rate of success of the use of a treatment based on radiofrequency for all the target stenosis. | 1 day
  Evaluation of the success of the use of bipolary radiofrequency for all target stenosis after each procedure

SECONDARY OUTCOMES:
Technic efficiency (Measure the duration of biliary permeability in the time) | From date of end of the treatment and the date of the first one re-permeabilisation of the prosthesis (until end of follow-up: 1 year)
  Ablation Therapy
Number of intervention for biliary drainage on the duration of the follow-up | From day of intervention until follow-up (during 1 year)
  Biliary drainage intervention
Global morbidity to 30 days | From day of intervention until 30 days
  Morbidity
Specific morbidity to 30 days | From day of intervention until 30 days
  Complications after intervention((cholecystitis, haemorrhage, pancreatitis, angiocholitis, intestinal perforation),
Overall survival | From day of intervention until 12 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: BORIES Erwan, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut Paoli-Calmettes — http://www.institutpaolicalmettes.fr